CLINICAL TRIAL: NCT05412992
Title: A Double-Blind, Placebo-Controlled Evaluation of the Dexmedetomidine Transdermal Systems for Postoperative Analgesia Following Abdominoplasty
Brief Title: Evaluation of the Dexmedetomidine Transdermal Systems for Postoperative Analgesia Following Abdominoplasty
Acronym: DMT2111
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: The SMC recommended stopping the trial. hemodynamic effects.
Sponsor: Teikoku Pharma USA, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: TPU-DMT-02-2111
Record Dates: First submitted 2022-06-01; First posted 2022-06-09 (Actual); Last update posted 2025-12-24 (Actual); Status verified 2025-12

CONDITIONS: Pain, Postoperative
Keywords: Abdominoplasty; Pain; Transdermal; DMTS
MeSH Terms: conditions — Pain, Postoperative; Pain

STUDY DESIGN:
Intervention Model Description: Subjects will be randomized in 1:1 ratio to receive DMTS or matching placebo
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: The sponsor, the investigator, personnel at the clinical study unit who are directly involved with monitoring and/or performing study procedures and assessments, and the subjects will be blinded to treatment assignment
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- DMTS Patch (Active Comparator): DMTS applied to upper outer arm
  Interventions: Drug: DMTS Patch
- Placebo Patch (Placebo Comparator): Placebo system (with no drug) to match DMTS applied to the upper arm
  Interventions: Drug: Placebo Patch

INTERVENTIONS:
Drug: DMTS Patch — DMTS applied before surgery and worn for 96 hours
  Other Names: DMTS
  Arms: DMTS Patch
Drug: Placebo Patch — Matching patches that have no active drug applied before surgery and worn for 96 hours
  Other Names: Placebo
  Arms: Placebo Patch

SUMMARY:
The primary objective of this study is to evaluate the analgesic efficacy of DMTS, compared with placebo, in subjects following abdominoplasty.

DETAILED DESCRIPTION:
This is a randomized, double-blind, placebo-controlled, one-time application study of DMTS or matching placebo over a 4-day treatment period (Day 1 Time 0 occurs when the DMTS or matching placebo systems have been applied). Subjects scheduled for an abdominoplasty will be screened up to 28 days prior to surgery. Eligible subjects will be randomized equally to treatment with DMTS or matching placebo. An independent safety monitoring committee will periodically review unblinded safety data to confirm the safety/tolerability of the dose or recommend a dose reduction.

ELIGIBILITY:
Inclusion Criteria:

* Male or female, ≥ 18 years of age.
* Scheduled to undergo a full abdominoplasty (including repair of small incidental abdominal hernias, but not including liposuction).
* Have a physical status classification of 1 or 2 per the American Society of Anesthesiology.
* Have a body weight > 58 kg, and body mass index of 20 to 38 kg/m2, inclusive.

Exclusion Criteria:

* Known sensitivity to dexmedetomidine or any excipient in the DMTS/placebo or to any peri- or postoperative medication whose use is required in this study.
* Skin abnormality (eg, scar, tattoo) or unhealthy skin condition (eg, burns, wounds) at the DMTS/matching placebo application site, according to examination by the investigator at screening or admission to the clinic prior to surgery.
* History of deep vein thrombosis or factor V Leiden deficiency.
* History of syncope or other syncopal attacks.
* Present and/or significant history of postural hypotension (determined through examination by the investigator or designee), or history of severe dizziness or fainting on standing in the opinion of the investigator.
* Evidence of a clinically significant 12-lead ECG abnormality.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 179 (Actual)
Dates: Start 2022-07-07 (Actual); Primary Completion 2023-04-19 (Actual); Study Completion 2023-04-19 (Actual)

PRIMARY OUTCOMES:
Time-interval weighted summed pain intensity (SPI) at designated time points | 5 to 96 hours following surgery
  The SPI measured using the 11-point (0 to 10) numeric rating scale, where 0 is equal to no pain and 10 is equal to worst pain

SECONDARY OUTCOMES:
Time-interval weighted summed pain intensity (SPI) over various time intervals | 5 to 96 hours following surgery
  The SPI measured using the 11-point (0 to 10) numeric rating scale, where 0 is equal to no pain and 10 is equal to worst pain, measured at rest over various time intervals
Rescue Medication | Up to 96 hours post surgery
  The proportion of subjects using rescue analgesic medication
Rescue Medication units | Up to 96 hours post surgery
  Total dose of rescue analgesic medication (in morphine-equivalent units)
Integrated Pain score and Rescue Medication | Up to 96 hours post surgery
  Integrated assessment of summed pain intensity (SPI) using the 11-point (0 to 10) numeric rating scale, where 0 is equal to no pain and 10 is equal to worst pain, at the time Rescue Medication was administered

CONTACTS AND LOCATIONS:
Overall Officials: James Song, MS, MA, Study Director — Teikoku Pharma USA, Inc.
Locations (2):
- United States (2):
  - Anaheim Clinical Trials, LLC, Anaheim, California
  - JBR Clinical Research, Salt Lake City, Utah

IPD SHARING:
Plan to Share IPD: No
No plan is in place to share individual participant data at this time.